CLINICAL TRIAL: NCT01337063
Title: Multi-Center Medication Reconciliation Quality Improvement Study
Acronym: MARQUIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Society of Hospital Medicine (Other); Vanderbilt University (Other); University of Wisconsin, Madison (Other); University of California, San Francisco (Other); Baystate Health (Other); University of Chicago (Other); Presbyterian Hospital, Charlotte (Unknown); Sioux Falls VA Health Care System (U.S. Federal Agency); Emory Johns Creek Hospital (Unknown)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P001814; 1R18HS019598 (AHRQ)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Adverse Drug Events; Medication Administered in Error
Keywords: Adverse drug events
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention (No Intervention): Usual care regarding medication reconciliation as currently practiced at each participating site.
- Intervention (Experimental): Improved medication reconciliation process using continuous quality improvement methods, mentored implementation, and an implementation guide.
  Interventions: Other: Mentored medication reconciliation quality improvement

INTERVENTIONS:
Other: Mentored medication reconciliation quality improvement — Based on expert recommendations from a recent conference on medication reconciliation sponsored by the Society of Hospital Medicine and funded by AHRQ, investigators will engage a steering committee and conduct a second conference to operationalize these recommendations into a set of "best practice" guidelines, standards, and tools to be adapted by each of 6 participating sites. After training mentors and developing data collection tools, a mentored quality improvement project will be conducted for 21 months, in which each site works to improve medication reconciliation using the toolkit and with mentorship in the form of two site visits and monthly phone calls.
  Arms: Intervention

SUMMARY:
Patients often have problems after they leave the hospital, in part because errors are made in the medications they are prescribed. The goal of this project is to develop a more accurate and safe medication prescription process when patients enter and leave the hospital and implement this process at six U.S. hospitals. The investigators will measure the success of the project and develop lessons learned so this process can be applied to other hospitals.

DETAILED DESCRIPTION:
Unintentional medication discrepancies during transitions in care (such as hospitalization and subsequent discharge) are very common and represent a major threat to patient safety. One solution to this problem is medication reconciliation. In response to Joint Commission requirements, most hospitals have developed medication reconciliation processes, but some have been more successful than others, and there are reports of pro-forma compliance without substantial improvements in patient safety. There is now collective experience about effective approaches to medication reconciliation, but these have yet to be consolidated, evaluated rigorously, and disseminated effectively.

This project's findings should provide valuable lessons to all hospitals regarding the best ways to design and implement medication reconciliation interventions to improve medication safety during transitions in care.

SPECIFIC AIMS:

Aim 1: Develop a toolkit consolidating the best practice recommendations for medication reconciliation

Aim 2: Conduct a multi-center mentored quality improvement project in which each site adapts the tools for its own environment and implements them

Aim 3: Assess the effects of a mentored medication reconciliation quality improvement intervention on unintentional medication discrepancies with potential for patient harm

Aim 4: Conduct rigorous program evaluation to determine the most important components of a medication reconciliation program and how best to implement it

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Admitted to inpatient medical or surgical services

Exclusion Criteria:

* Vulnerable populations (pregnant women, prisoners, institutionalized individuals)
* Under 18 years

Hospital staff subjects:

* Personnel directly involved in the medication reconciliation process, which depending on the site might include residents, physician assistants, inpatient attending physicians, nurses, pharmacists, and pharmacy technicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1836 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be unintentional medication discrepancies in admission orders and discharge orders with potential for patient harm | 6 months prior to implementation of intervention to 21 months during intervention
  The primary outcome will be determined by a study pharmacist who will take a "gold standard" medication history on 5 patients per week, then compare that history to the medical team's medication history, to admission orders, and to discharge orders. Any unintentional medication discrepancies in orders will be recorded. A physician adjudicator will then make a final determination regarding whether an error occurred, the type of error, the potential for patient harm, and the potential severity.

SECONDARY OUTCOMES:
Patient satisfaction | 6 months prior to implementation of intervention to 21 months during intervention
  Patient Satisfaction will be assessed using data from the HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) survey. This survey is already administered to a sample of patients from all hospitals; we will measure both global satisfaction and questions related to medications (e.g., "before giving you any new medications, how often did hospital staff tell you what the medicine was for," and "before giving you any new medications, how often did hospital staff describe possible site effects in a way you could understand.")
Administrative outcomes | 6 months prior to implementation of intervention to 21 months during intervention
  Emergency Department (ED) or hospital readmission to the same institution within 30 days of discharge, using computerized hospital records of all eligible patients.
Total medication discrepancies | 6 months prior to implementation of intervention to 21 months during intervention
  As with Outcome 1, but without adjudication for potential for harm

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - University of Chicago Hospitals and Clinics, Chicago, Illinois
  - Baystate Health, Springfield, Massachusetts
  - Presbyterian Hospital, Charlotte, North Carolina
  - Sioux Falls VA Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Background] Coleman EA, Smith JD, Raha D, Min SJ. Posthospital medication discrepancies: prevalence and contributing factors. Arch Intern Med. 2005 Sep 12;165(16):1842-7. doi: 10.1001/archinte.165.16.1842. PMID 16157827
- [Background] Cornish PL, Knowles SR, Marchesano R, Tam V, Shadowitz S, Juurlink DN, Etchells EE. Unintended medication discrepancies at the time of hospital admission. Arch Intern Med. 2005 Feb 28;165(4):424-9. doi: 10.1001/archinte.165.4.424. PMID 15738372
- [Background] Schnipper JL, Kirwin JL, Cotugno MC, Wahlstrom SA, Brown BA, Tarvin E, Kachalia A, Horng M, Roy CL, McKean SC, Bates DW. Role of pharmacist counseling in preventing adverse drug events after hospitalization. Arch Intern Med. 2006 Mar 13;166(5):565-71. doi: 10.1001/archinte.166.5.565. PMID 16534045
- [Background] Institute for Healthcare Improvement. Medication Reconciliation Review. 2007; http://www.ihi.org/IHI/Topics/PatientSafety/MedicationSystems/Tools/Medication+Reconciliation+Review.htm. Accessed January 7, 2010.
- [Background] Tam VC, Knowles SR, Cornish PL, Fine N, Marchesano R, Etchells EE. Frequency, type and clinical importance of medication history errors at admission to hospital: a systematic review. CMAJ. 2005 Aug 30;173(5):510-5. doi: 10.1503/cmaj.045311. PMID 16129874
- [Background] Pippins JR, Gandhi TK, Hamann C, Ndumele CD, Labonville SA, Diedrichsen EK, Carty MG, Karson AS, Bhan I, Coley CM, Liang CL, Turchin A, McCarthy PC, Schnipper JL. Classifying and predicting errors of inpatient medication reconciliation. J Gen Intern Med. 2008 Sep;23(9):1414-22. doi: 10.1007/s11606-008-0687-9. Epub 2008 Jun 19. PMID 18563493
- [Background] Vira T, Colquhoun M, Etchells E. Reconcilable differences: correcting medication errors at hospital admission and discharge. Qual Saf Health Care. 2006 Apr;15(2):122-6. doi: 10.1136/qshc.2005.015347. PMID 16585113
- [Background] Wortman SB. Medication reconciliation in a community, nonteaching hospital. Am J Health Syst Pharm. 2008 Nov 1;65(21):2047-54. doi: 10.2146/ajhp080091. PMID 18945865
- [Background] Schnipper JL, Hamann C, Ndumele CD, Liang CL, Carty MG, Karson AS, Bhan I, Coley CM, Poon E, Turchin A, Labonville SA, Diedrichsen EK, Lipsitz S, Broverman CA, McCarthy P, Gandhi TK. Effect of an electronic medication reconciliation application and process redesign on potential adverse drug events: a cluster-randomized trial. Arch Intern Med. 2009 Apr 27;169(8):771-80. doi: 10.1001/archinternmed.2009.51. PMID 19398689
- [Background] Doyle E. Medication reconciliation done right. Today's Hospitalist. September 2009.
- [Background] Coffey M, Cornish P, Koonthanam T, Etchells E, Matlow A. Implementation of admission medication reconciliation at two academic health sciences centres: challenges and success factors. Healthc Q. 2009;12 Spec No Patient:102-9. doi: 10.12927/hcq.2009.20719. PMID 19667786
- [Background] Brown C, Lilford R. Evaluating service delivery interventions to enhance patient safety. BMJ. 2008 Dec 17;337:a2764. doi: 10.1136/bmj.a2764. No abstract available. PMID 19091764
- [Background] Schnipper JL, Roumie CL, Cawthon C, Businger A, Dalal AK, Mugalla I, Eden S, Jacobson TA, Rask KJ, Vaccarino V, Gandhi TK, Bates DW, Johnson DC, Labonville S, Gregory D, Kripalani S; PILL-CVD Study Group. Rationale and design of the Pharmacist Intervention for Low Literacy in Cardiovascular Disease (PILL-CVD) study. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):212-9. doi: 10.1161/CIRCOUTCOMES.109.921833. PMID 20233982
- [Background] Agency for Healthcare Research and Quality. CAHPS Hospital Survey (H-CAHPS) 2009; https://www.cahps.ahrq.gov/content/products/HOSP/PROD_HOSP_Intro.asp?p=1022&s=221. Accessed January 15, 2010.
- [Background] Parry C, Mahoney E, Chalmers SA, Coleman EA. Assessing the quality of transitional care: further applications of the care transitions measure. Med Care. 2008 Mar;46(3):317-22. doi: 10.1097/MLR.0b013e3181589bdc. PMID 18388847
- [Background] Kivimaki M, Elovainio M. A short version of the Team Climate Inventory: development and psychometric properties. Journal of Occupational and Organizational Psychology. 1999;72:241-246.
- [Background] Cochrane Collaboration. Effective Practice and Organization of Care (EPOC) Methods Paper: Including interrupted time series (ITS) designs in a EPOC review. 1998.
- [Background] Bazeley P. Computerized data analysis for mixed methods research. In: Tashakkori A, Teddlie C, eds. Mixed methodology: combining qualitative and quantitative approaches. Thousand Oaks, CA: Sage; 2003.
- [Background] Glasser B, Strauss A. Discovery of grounded theory: strategies for qualitative research. Chicago: Adeline; 1967.
- [Background] Strauss A, Corbin. Basics of qualitative research: grounded theory procedures and techniques. 2nd ed. Thousand Oaks, CA: Sage; 1998.
- [Background] Patton MQ. Qualitative research & evaluation methods. 3rd ed. Thousand Oaks, CA: Sage; 2002.
- [Background] Miles M, Huberman AM. Qualitative data analysis: an expanded sourcebook. 2nd ed. Newbury Park, CA: Sage; 1994.
- [Background] Dumas JE, Lynch AM, Laughlin JE, Phillips Smith E, Prinz RJ. Promoting intervention fidelity. Conceptual issues, methods, and preliminary results from the EARLY ALLIANCE prevention trial. Am J Prev Med. 2001 Jan;20(1 Suppl):38-47. doi: 10.1016/s0749-3797(00)00272-5. PMID 11146259
- [Background] Joint Commission on Accreditation of Healthcare Organizations. Joint Commission Fact Sheets: Facts about the tracer methodology. 2006; http://www.jointcommission.org/AboutUs/Fact_Sheets/Tracer_Methodology.htm. Accessed January 15, 2010.
- [Background] Agency for Healthcare Research and Quality. Hospital Survey on Patient Safety Culture. 2009; http://www.ahrq.gov/qual/patientsafetyculture/hospsurvindex.htm. Accessed January 10, 2010.
- [Background] Joint Commission on Accreditation of Healthcare Organizations. Accreditation Program: Hospital 2011 National Patient Safety Goals; http://www.jointcommission.org/assets/1/6/2011_NPSGs_HAP.pdf. Accessed April 12, 2011.
- [Background] Gillespie U, Alassaad A, Henrohn D, Garmo H, Hammarlund-Udenaes M, Toss H, Kettis-Lindblad A, Melhus H, Morlin C. A comprehensive pharmacist intervention to reduce morbidity in patients 80 years or older: a randomized controlled trial. Arch Intern Med. 2009 May 11;169(9):894-900. doi: 10.1001/archinternmed.2009.71. PMID 19433702
- [Background] Koehler BE, Richter KM, Youngblood L, Cohen BA, Prengler ID, Cheng D, Masica AL. Reduction of 30-day postdischarge hospital readmission or emergency department (ED) visit rates in high-risk elderly medical patients through delivery of a targeted care bundle. J Hosp Med. 2009 Apr;4(4):211-8. doi: 10.1002/jhm.427. PMID 19388074
- [Background] Midlov P, Deierborg E, Holmdahl L, Hoglund P, Eriksson T. Clinical outcomes from the use of Medication Report when elderly patients are discharged from hospital. Pharm World Sci. 2008 Dec;30(6):840-5. doi: 10.1007/s11096-008-9236-1. Epub 2008 Jul 25. PMID 18654837
- [Derived] Mixon AS, Kripalani S, Stein J, Wetterneck TB, Kaboli P, Mueller S, Burdick E, Nolido NV, Labonville S, Minahan JA, Orav EJ, Goldstein J, Schnipper JL. An On-Treatment Analysis of the MARQUIS Study: Interventions to Improve Inpatient Medication Reconciliation. J Hosp Med. 2019 Oct 1;14(10):614-617. doi: 10.12788/jhm.3308. Epub 2019 Aug 16. PMID 31433768
- [Derived] Schnipper JL, Mixon A, Stein J, Wetterneck TB, Kaboli PJ, Mueller S, Labonville S, Minahan JA, Burdick E, Orav EJ, Goldstein J, Nolido NV, Kripalani S. Effects of a multifaceted medication reconciliation quality improvement intervention on patient safety: final results of the MARQUIS study. BMJ Qual Saf. 2018 Dec;27(12):954-964. doi: 10.1136/bmjqs-2018-008233. Epub 2018 Aug 20. PMID 30126891
- [Derived] Salanitro AH, Kripalani S, Resnic J, Mueller SK, Wetterneck TB, Haynes KT, Stein J, Kaboli PJ, Labonville S, Etchells E, Cobaugh DJ, Hanson D, Greenwald JL, Williams MV, Schnipper JL. Rationale and design of the Multicenter Medication Reconciliation Quality Improvement Study (MARQUIS). BMC Health Serv Res. 2013 Jun 25;13:230. doi: 10.1186/1472-6963-13-230. PMID 23800355